CLINICAL TRIAL: NCT00294970
Title: Cognitive Characteristics of PTSD Patients With OCD
Status: Completed | Type: Observational
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Prof. Joseph Zohar, Chaim Sheba Medical Center
Other Study IDs: SHEBA-05-3918-JZ-CTIL
Record Dates: First submitted 2006-02-19; First posted 2006-02-22 (Estimated); Last update posted 2010-02-02 (Estimated); Status verified 2010-01

CONDITIONS: Post-Traumatic Stress Disorders; Obsessive-Compulsive Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Obsessive-Compulsive Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- PTSD: Patients with diagnosis of PTSD
- OCD: Patients with diagnosis of OCD
- PTSD/OCD: Patients with diagnosis of comorbid PTSD and OCD

SUMMARY:
Cognitive profile of patients who suffer both from PTSD and OCD, as compared to those who suffer from PTSD or OCD without other comorbidity.

DETAILED DESCRIPTION:
Demographic data and cognitive data will be compared on PTSD, PTSD-OCD and OCD patients using a battery of computerized cognitive tests

ELIGIBILITY:
Inclusion Criteria:

* Patients suffer from current PTSD with no other co-morbidity
* Patients suffer from current OCD with no other co-morbidity
* Patients suffer from current PTSD and OCD

Exclusion Criteria:

* Patients suffer from PTSD and OC symptoms

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients from each group were invited to participate in the study from the inpatient, outpatient and public clinic populations of the Chaim Sheba Medical Center Psychiatric Division
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2006-02; Study Completion 2006-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Zohar, MD, Study Director — Sheba Medical Center
Locations (1):
- Chaim Sheba Medical Center, Ramat Gan, Israel